CLINICAL TRIAL: NCT02626546
Title: Predictors, Risk Factors and Outcome Following Major Surgery
Acronym: PROFS
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: Norrlands University Hospital (Other); Region Örebro County (Other); University Hospital, Linkoeping (Other); Uppsala University Hospital (Other)
Responsible Party: Principal Investigator, Sigridur Kalman, Medical doctor, PHD, Karolinska Institutet
Other Study IDs: 2015/1128-31/4
Record Dates: First submitted 2015-11-06; First posted 2015-12-10 (Estimated); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Surgical Procedure, Unspecified; Postoperative Complications
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Major surgical procedures: All patients selected to follow up
  Interventions: Procedure: Major surgical procedure

INTERVENTIONS:
Procedure: Major surgical procedure — observation of postoperative outcomes

SUMMARY:
This is a multicentre, prospective, observational cohort study. Consecutive patients, operated in six University Hospitals in Sweden will be recruited following major surgical procedure. The length of patient recruitment period will be 12 weeks. The length of follow up will be 360 days . The objectives are to determine the postoperative morbidity (during the hospital stay), the survival (0-360 days), to identify risk factors for adverse outcomes and to identify risk factors that may potentially be influenced by any intervention in the future.

Amendments:

1. The follow-up of mortality is extended to 3 years of the cohort
2. The mortality of the background population at 30 and 90 Days will be analyzed
3. Validation of the Surgical Outcome Risk Tool in the study cohort and in the background population are planned

DETAILED DESCRIPTION:
This is a multicenter, prospective, observational study. Length of patient recruitment is 12 weeks, the length of observation is 360 postoperative days. The expected number of patients is 1000.

Patients will be selected from the operation planning software on each study site. It is done by daily screening of the operation list and will be enrolled by applying the inclusion criteria. The criteria of surgical severity will be assessed by the UK surgical severity grading system ( AXA PPP/ Specialist Procedure Codes, United Kingdom). For that purpose a scroll list will be used, which is available on the website of the Surgical Outcome Risk Tool calculator.

Patient characteristics will be prospectively collected from medical records: age, gender, co-morbidities, medical history, physical activity, blood pressure, heart rate, oxygen saturation and neurological function; routine laboratory findings; type, complexity, urgency of surgery, incision localization and malignancy; lowest intraoperative systolic blood pressure, heart rate. The outcomes are the postoperative morbidity (assessed by the Postoperative Morbidity Survey) classified by the Clavien-Dindo classification tool (during hospital stay), and mortality, use of medications, hospital re-admissions (0-360 days) and new occurrence in different disease related national quality registries.Relationships between postoperative morbidity (POMS) the severity of morbidity (Clavien Dindo) and mortality will be analyzed. For illustration, Kaplan Meyer plots will be used, and for analyses Cox proportional hazard model will be used with adjustment for sex and age.

Additional changes:

1. The length of observation for survival was extended to 3 years. The mortality at 3 years will be analyzed addressing the relationship between the postoperative morbidity (POMS) and mortality. Cox regression model will be used with adjustment of age, comorbidity and malignancy.
2. Validation of Surgical Outcome Risk Tool is planned in two populations related to the PROFS study: eligible and background population. As the PROFS cohort was manually selected, we presumed that the eligible population is larger than the enrolled population.To enable electronic selection of the eligible population, we have developed a script, which translates the Swedish surgical codes into the UK severity codes. Using the same script we will classify the surgical severity in the background population of the PROFS cohort. Variables included in the Surgical Outcome Risk Tool will be extracted from the operation databases of each study site. The date of death will be extracted from the Swedish National Adress Registry and the malignancy from the registry of National Swedish Cancer Registry.

ELIGIBILITY:
Eligibility Criteria:

Sex: male or female Age limits: minimum age 18 Years maximum age: no limits

Inclusion criteria:

* individuals classified by the American Society of Anesthesiologists Physical Status Classification System (ASA) ≥ 3 AND
* are scheduled for elective or emergency surgical procedure classified as -major OR major/complex by Surgical Outcome Risk Tool (SORT)

Non eligibility criteria are the following surgical procedures:

* organ transplantation
* immediate trauma
* breast
* ear, nose throat
* central nervous system
* cardiac, vascular, pulmonary,
* face, mouth, salivary, thyroidea
* skin, subcutaneous tissue
* endoscopic gastrointestinal
* lack of Swedish identity number

Exclusion Criteria:

* patients who refuse the follow up
* patients who are not available for the follow up (living in other countries)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive adult patients who are operated for major surgical procedures during the study period in tertiary hospitals in Sweden.
Sampling Method: Non-Probability Sample
Enrollment: 1061 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2020-09 (Actual)

PRIMARY OUTCOMES:
postoperative complications | 3-10 postoperative days
  postoperative morbidity survey, Clavien Dindo

SECONDARY OUTCOMES:
postoperative mortality | 30-360 postoperative days and 3 years
  number of deaths at 30, 360 Days AND 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Sigriduar Kalman, MD PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska University Hospital, Huddinge, Sweden